CLINICAL TRIAL: NCT02057250
Title: A Multicenter, Randomized, Open-Label, Parallel-Group Usability Study Of The Sarilumab Auto-Injector Device And A Prefilled Syringe In Patients With Moderate To Severe Active Rheumatoid Arthritis Who Are Candidates For Anti-IL6R Therapy
Brief Title: To Evaluate Sarilumab - SAR153191 (REGN88) - Auto-injector Device In Patients With Rheumatoid Arthritis
Acronym: SARIL-RA-EASY
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MSC12665; 2012-004339-21; U1111-1130-9931 (Other: UTN)
Record Dates: First submitted 2014-01-31; First posted 2014-02-07 (Estimated); Results first posted 2017-06-20 (Actual); Last update posted 2017-06-20 (Actual); Status verified 2017-05

CONDITIONS: RA
MeSH Terms: interventions — sarilumab; Methotrexate; Sulfasalazine; Leflunomide; Hydroxychloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Sarilumab 150 mg by AID (Experimental): Sarilumab 150 mg subcutaneous (SC) injection every 2 weeks (q2w) administered by AID with one or a combination of non-biologic disease-modifying anti-rheumatic drug (DMARD) (hydroxychloroquine, methotrexate, sulfasalazine and/or Leflunomide, except for simultaneous combination use of leflunomide and methotrexate) in AID assessment phase for 12 weeks. Participants who completed 12 weeks AID assessment phase entered in open-label extension phase and received sarilumab 150 mg SC injection q2w administered by PFS with one or a combination of non-biologic DMARD for 52 weeks.
  Interventions: Drug: Sarilumab; Device: Auto-Injector Device (AID); Drug: Methotrexate; Drug: Sulfasalazine; Drug: Leflunomide; Drug: Hydroxychloroquine
- Sarilumab 150 mg by PFS (Experimental): Sarilumab 150 mg SC injection q2w administered by PFS with one or a combination of non-biologic DMARD (hydroxychloroquine, methotrexate, sulfasalazine and/or Leflunomide, except for simultaneous combination use of leflunomide and methotrexate) in AID assessment phase for 12 weeks. Participants who completed 12 weeks AID assessment phase entered in open-label extension phase and received sarilumab 150 mg SC injection q2w administered by PFS with one or a combination of non-biologic DMARD for 52 weeks.
  Interventions: Drug: Sarilumab; Device: Pre-filled Syringe (PFS); Drug: Methotrexate; Drug: Sulfasalazine; Drug: Leflunomide; Drug: Hydroxychloroquine
- Sarilumab 200 mg by AID (Experimental): Sarilumab 200 mg SC injection q2w administered by AID with one or a combination of non-biologic DMARD (hydroxychloroquine, methotrexate, sulfasalazine and/or Leflunomide, except for simultaneous combination use of leflunomide and methotrexate) in AID assessment phase for 12 weeks. Participants who completed 12 weeks AID assessment phase entered in open-label extension phase and received sarilumab 150 mg SC injection q2w administered by PFS with one or a combination of non-biologic DMARD for 52 weeks.
  Interventions: Drug: Sarilumab; Device: Auto-Injector Device (AID); Drug: Methotrexate; Drug: Sulfasalazine; Drug: Leflunomide; Drug: Hydroxychloroquine
- Sarilumab 200 mg by PFS (Experimental): Sarilumab 200 mg SC injection q2w administered by PFS with one or a combination of non-biologic DMARD (hydroxychloroquine, methotrexate, sulfasalazine and/or Leflunomide, except for simultaneous combination use of leflunomide and methotrexate) in AID assessment phase for 12 weeks. Participants who completed 12 weeks AID assessment phase entered in open-label extension phase and received sarilumab 150 mg SC injection q2w administered by PFS with one or a combination of non-biologic DMARD for 52 weeks.
  Interventions: Drug: Sarilumab; Device: Pre-filled Syringe (PFS); Drug: Methotrexate; Drug: Sulfasalazine; Drug: Leflunomide; Drug: Hydroxychloroquine

INTERVENTIONS:
Drug: Sarilumab — Pharmaceutical form: Solution Route of administration: Subcutaneous
  Other Names: SAR153191; REGN88
Device: Auto-Injector Device (AID)
  Arms: Sarilumab 150 mg by AID; Sarilumab 200 mg by AID
Device: Pre-filled Syringe (PFS)
  Arms: Sarilumab 150 mg by PFS; Sarilumab 200 mg by PFS
Drug: Methotrexate — Dispensed according to local practice.
Drug: Sulfasalazine — Dispensed according to local practice.
Drug: Leflunomide — Dispensed according to local practice.
Drug: Hydroxychloroquine — Dispensed according to local practice.

SUMMARY:
Primary Objective:

To collect real-use data of the sarilumab auto-injector device (AID) used by rheumatoid arthritis (RA) participants.

Secondary Objective:

To compare the pharmacokinetic (PK) exposure of sarilumab administered by AID versus prefilled syringes (PFS).

DETAILED DESCRIPTION:
Total study duration up to 74 weeks: screening up to 4 weeks, AID assessment phase of 12 weeks, extension phase of 52 weeks and post-treatment follow-up of 6 weeks.

For participants not entering the extension phase, total study duration up to 22 weeks (screening, AID assessment phase and follow-up).

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of RA, ≥3 months disease duration;
* Participant willing and able to self-inject;
* Continuous treatment with 1 or a combination of non-biologic disease modifying antirheumatic drugs (DMARDs) (except leflunomide in combination with methotrexate);
* Moderate-to-severely active RA.

Exclusion criteria:

* Participants <18 years;
* Prior treatment with anti-interleukin 6 (IL-6) or IL-6 receptor (IL-6R) antagonists;
* Treatment with tumor necrosis factor (TNF) antagonists;
* Treatment with RA-directed biologic agents other than with a TNF-α antagonist mechanism as follows: Anakinra, Abatacept, Rituximab or other cell-depleting agent;
* Prior treatment with a Janus kinase inhibitor.

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 217 (Actual)
Dates: Start 2014-03; Primary Completion 2015-02 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (53):
- United States (31):
  - Investigational Site Number 840152, Huntsville, Alabama
  - Investigational Site Number 840221, Peoria, Arizona
  - Investigational Site Number 840226, Roseville, California
  - Investigational Site Number 840223, Boulder, Colorado
  - Investigational Site Number 840229, Miami, Florida
  - Investigational Site Number 840236, Orlando, Florida
  - Investigational Site Number 840155, Palm Harbor, Florida
  - Investigational Site Number 840220, South Miami, Florida
  - Investigational Site Number 840202, Hagerstown, Maryland
  - Investigational Site Number 840232, Flint, Michigan
  - Investigational Site Number 840233, Kalamazoo, Michigan
  - Investigational Site Number 840037, Tupelo, Mississippi
  - Investigational Site Number 840112, Lincoln, Nebraska
  - Investigational Site Number 840039, Albany, New York
  - Investigational Site Number 840224, Cincinnati, Ohio
  - Investigational Site Number 840002, Oklahoma City, Oklahoma
  - Investigational Site Number 840065, Tulsa, Oklahoma
  - Investigational Site Number 840009, Duncansville, Pennsylvania
  - Investigational Site Number 840062, Reading, Pennsylvania
  - Investigational Site Number 840016, North Charleston, South Carolina
  - Investigational Site Number 840025, Jackson, Tennessee
  - Investigational Site Number 840038, Austin, Texas
  - Investigational Site Number 840230, Carrollton, Texas
  - Investigational Site Number 840001, Dallas, Texas
  - Investigational Site Number 840020, Houston, Texas
  - Investigational Site Number 840239, Houston, Texas
  - Investigational Site Number 840241, Houston, Texas
  - Investigational Site Number 840242, Houston, Texas
  - Investigational Site Number 840069, Lubbock, Texas
  - Investigational Site Number 840074, Mesquite, Texas
  - Investigational Site Number 840237, Plano, Texas
- Chile (4):
  - Investigational Site Number 152005, Osorno
  - Investigational Site Number 152050, Santiago
  - Investigational Site Number 152014, Talca
  - Investigational Site Number 152007, Viña del Mar
- Mexico (3):
  - Investigational Site Number 484002, Guadalajara
  - Investigational Site Number 484004, Mérida
  - Investigational Site Number 484005, Monterrey
- Poland (5):
  - Investigational Site Number 616002, Bialystok
  - Investigational Site Number 616005, Lublin
  - Investigational Site Number 616004, Warsaw
  - Investigational Site Number 616017, Warsaw
  - Investigational Site Number 616012, Wroclaw
- Russia (4):
  - Investigational Site Number 643006, Kemerovo
  - Investigational Site Number 643020, Moscow
  - Investigational Site Number 643001, Moscow
  - Investigational Site Number 643008, Saint Petersburg
- South Africa (6):
  - Investigational Site Number 710050, Bellville
  - Investigational Site Number 710011, Cape Town
  - Investigational Site Number 710007, Cape Town
  - Investigational Site Number 710003, Durban
  - Investigational Site Number 710001, Johannesburg
  - Investigational Site Number 710051, Port Elizabeth

REFERENCES:
- [Derived] Kivitz A, Baret-Cormel L, van Hoogstraten H, Wang S, Parrino J, Xu C, Stanislav M. Usability and Patient Preference Phase 3 Study of the Sarilumab Pen in Patients with Active Moderate-to-Severe Rheumatoid Arthritis. Rheumatol Ther. 2018 Jun;5(1):231-242. doi: 10.1007/s40744-017-0090-2. Epub 2017 Dec 5. PMID 29209946

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 53 centers in 6 countries. A total of 419 participants were screened between 18 March 2014 and 14 October 2014, out of which 217 participants were enrolled and treated.
Pre-assignment Details: Participants were randomized in 1:1:1:1 ratio to Sarilumab 150 mg administered by auto-injector device (AID) or prefilled syringe (PFS) or Sarilumab 200 mg administered by AID or PFS. Participants who completed 12-week AID assessment phase, were treated in open-label extension phase for 52 weeks.
Groups:
- Sarilumab 150 mg by AID (AID Assessment Phase): Sarilumab 150 mg subcutaneous (SC) injection every 2 weeks (q2w) administered by AID with one or a combination of non-biologic disease-modifying anti-rheumatic drug (DMARD) for 12 weeks.
- Sarilumab 150 mg by PFS (AID Assessment Phase): Sarilumab 150 mg SC injection q2w administered by PFS with one or a combination of non-biologic DMARD for 12 weeks.
- Sarilumab 200 mg by AID (AID Assessment Phase): Sarilumab 200 mg SC injection q2w administered by AID with one or a combination of non-biologic DMARD for 12 weeks.
- Sarilumab 200 mg by PFS (AID Assessment Phase): Sarilumab 200 mg SC injection q2w administered by PFS with one or a combination of non-biologic DMARD for 12 weeks.
- Sarilumab 150 mg by PFS (Extension Phase): Participants who completed 12 week AID assessment phase received Sarilumab 150 mg SC injection q2w administered by PFS with one or a combination of non-biologic DMARD for 52 weeks.
Period: AID Assessment Phase
Arm/Group | Sarilumab 150 mg by AID (AID Assessment Phase) | Sarilumab 150 mg by PFS (AID Assessment Phase) | Sarilumab 200 mg by AID (AID Assessment Phase) | Sarilumab 200 mg by PFS (AID Assessment Phase) | Sarilumab 150 mg by PFS (Extension Phase)
Started | 56 | 53 | 52 | 56 | 0
Completed | 52 | 50 | 45 | 54 | 0
Not Completed | 4 | 3 | 7 | 2 | 0
Not completed — Adverse Event | 3 | 2 | 6 | 1 | 0
Not completed — Other than specified above | 1 | 1 | 1 | 1 | 0
Period: Extension Phase
Arm/Group | Sarilumab 150 mg by AID (AID Assessment Phase) | Sarilumab 150 mg by PFS (AID Assessment Phase) | Sarilumab 200 mg by AID (AID Assessment Phase) | Sarilumab 200 mg by PFS (AID Assessment Phase) | Sarilumab 150 mg by PFS (Extension Phase)
Started | 0 | 0 | 0 | 0 | 192 (9 participants who completed AID Assessment phase did not enter extension phase.)
Treated | 0 | 0 | 0 | 0 | 188
Completed | 0 | 0 | 0 | 0 | 156
Not Completed | 0 | 0 | 0 | 0 | 36
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 15
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 10
Not completed — Entered in this period but not treated | 0 | 0 | 0 | 0 | 4
Not completed — Other than specified above | 0 | 0 | 0 | 0 | 7

BASELINE CHARACTERISTICS:
Groups:
- Sarilumab 150 mg by AID (AID Assessment Phase): Sarilumab 150 mg SC injection q2w administered by AID with one or a combination of non-biologic DMARD for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Sarilumab 150 mg by AID (AID Assessment Phase) | Sarilumab 150 mg by PFS (AID Assessment Phase) | Sarilumab 200 mg by AID (AID Assessment Phase) | Sarilumab 200 mg by PFS (AID Assessment Phase) | Total
Number analyzed (Participants) | 56 | 53 | 52 | 56 | 217
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.7 (13.8) | 54.2 (14.2) | 55.9 (12.3) | 50.3 (12.8) | 53.5 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 43 | 44 | 49 | 181
  Male | 11 | 10 | 8 | 7 | 36

OUTCOME MEASURES:

1. Primary Outcome: Number of Validated AID Associated Product Technical Failures (PTFs)
Description: A PTF was defined as any product technical complaint (PTC) related to the use of the AID that had a validated technical cause. Each participant was given a diary having questions related to participant's ability to remove the cap, to start the injection, to complete the injection and regarding confirmation of completing the injection. Participants were asked to answer the questions each time they self-inject the sarilumab. If the response was "no" to any of the first 3 questions, this was considered as a PTC. The used AID, for which PTC was reported, was sent to sponsor, examined and evaluated for the occurrence of a PTF.
Time Frame: Baseline up to Week 12
Population: Modified intent-to-treat (mITT) population included all randomized participants who received at least 1 dose of investigational medicinal product (IMP) with AID and attended at least 1 post-baseline visit during AID assessment phase of the study.
Measure: Number; unit: PTFs
Units Other Than Participants: Injections
Arm/Group | Sarilumab 150 mg by AID (AID Assessment Phase) | Sarilumab 200 mg by AID (AID Assessment Phase)
Number analyzed (Participants) | 56 | 52
Number analyzed (Injections) | 312 | 288
PTFs | 0 | 0

2. Secondary Outcome: Area Under the Serum Concentration Versus Time Curve Calculated Using the Trapezoidal Method During a Dose Interval (AUC[0-tau]) for Sarilumab
Description: AUC(0-tau) is defined as area under the serum concentration versus time curve calculated using the trapezoidal method during a dose interval, where dose interval was 2 weeks. Serum concentrations of sarilumab were analyzed using validated enzyme linked immunosorbent assay (ELISA).
Time Frame: Week 0-2: pre-dose on Day 1, anytime post-dose on Day 3, Day 5, Day 8, Day 12, Day 15; Week 10-12: pre-dose on Day 71, anytime post-dose on Day 73, Day 75, Day 78, Day 82, Day 85
Population: Pharmacokinetic(PK) population included all randomized participants who received at least 1 dose of IMP and have least 1 PK parameter calculated using non compartmental methods following the first (Day 1) or sixth administration (Day 71). Here, Number Analyzed = participants with available data for specified category for each arm, respectively.
Measure: Mean (Standard Deviation); unit: mg*day/L
Arm/Group | Sarilumab 150 mg by AID (AID Assessment Phase) | Sarilumab 150 mg by PFS (AID Assessment Phase) | Sarilumab 200 mg by AID (AID Assessment Phase) | Sarilumab 200 mg by PFS (AID Assessment Phase)
Number analyzed (Participants) | 56 | 53 | 52 | 56
mg*day/L
  Week 0-2: number analyzed (Participants) | 39 | 34 | 34 | 41
  Week 0-2 | 131 (54.5) | 152 (76.7) | 235 (117) | 227 (94.9)
  Week 10-12: number analyzed (Participants) | 44 | 40 | 36 | 38
  Week 10-12 | 205 (126) | 220 (130) | 455 (294) | 405 (244)

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs) were collected from signature of the informed consent form up to the final visit (74 Weeks) regardless of seriousness or relationship to study drug.
Description: Reported AEs are treatment-emergent AEs developed/worsened during 'on treatment period' (time from first dose of IMP in AID assessment phase up to last dose of IMP in extension phase + 6 weeks). Safety population of AID assessment phase included all randomized participants who received at least 1 dose or part of a dose of IMP and safety population of extension phase included all participants who continued in the extension phase and received at least 1 dose or part of a dose of IMP.
Arm/Group | Sarilumab 150 mg by AID (AID Assessment Phase) | Sarilumab 150 mg by PFS (AID Assessment Phase) | Sarilumab 200 mg by AID (AID Assessment Phase) | Sarilumab 200 mg by PFS (AID Assessment Phase) | Sarilumab 150 mg by PFS (Extension Phase)
Serious Adverse Events (participants affected / at risk) | 1/56 | 0/53 | 3/52 | 4/56 | 19/188
Other Adverse Events (participants affected / at risk) | 29/56 | 21/53 | 24/52 | 23/56 | 83/188
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sarilumab 150 mg by AID (AID Assessment Phase) (N=56) | Sarilumab 150 mg by PFS (AID Assessment Phase) (N=53) | Sarilumab 200 mg by AID (AID Assessment Phase) (N=52) | Sarilumab 200 mg by PFS (AID Assessment Phase) (N=56) | Sarilumab 150 mg by PFS (Extension Phase) (N=188)
Bursitis infective staphylococcal (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Erysipelas (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Vertebrobasilar insufficiency (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 1
Coronary artery occlusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Wolff-Parkinson-White syndrome (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Thrombophlebitis superficial (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Rheumatoid lung (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Traumatic arthritis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sarilumab 150 mg by AID (AID Assessment Phase) (N=56) | Sarilumab 150 mg by PFS (AID Assessment Phase) (N=53) | Sarilumab 200 mg by AID (AID Assessment Phase) (N=52) | Sarilumab 200 mg by PFS (AID Assessment Phase) (N=56) | Sarilumab 150 mg by PFS (Extension Phase) (N=188)
Bronchitis (Infections and infestations) | 4 | 1 | 1 | 1 | 8
Nasopharyngitis (Infections and infestations) | 4 | 1 | 1 | 2 | 4
Pharyngitis (Infections and infestations) | 5 | 0 | 1 | 1 | 2
Sinusitis (Infections and infestations) | 1 | 3 | 0 | 1 | 12
Upper respiratory tract infection (Infections and infestations) | 3 | 2 | 1 | 3 | 25
Urinary tract infection (Infections and infestations) | 2 | 2 | 2 | 2 | 10
Leukopenia (Blood and lymphatic system disorders) | 3 | 2 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 10 | 9 | 6 | 4 | 12
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 1 | 2 | 1 | 3
Hypertension (Vascular disorders) | 2 | 1 | 3 | 2 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 3 | 0
Injection site erythema (General disorders) | 2 | 2 | 4 | 4 | 7
Injection site pruritus (General disorders) | 1 | 2 | 0 | 4 | 5
Alanine aminotransferase increased (Investigations) | 1 | 1 | 5 | 1 | 9
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 3 | 8
Contusion (Injury, poisoning and procedural complications) | 3 | 0 | 0 | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.